CLINICAL TRIAL: NCT01035450
Title: Randomized Evaluation of Sirolimus-eluting Versus Everolimus-eluting Stent Trial
Acronym: RESET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C338
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus-eluting stent (Experimental)
  Interventions: Device: Everolimus-eluting stent
- Sirolimus-eluting stent (Active Comparator)
  Interventions: Device: Sirolimus-eluting stent

INTERVENTIONS:
Device: Everolimus-eluting stent — Everolimus-eluting stent
  Arms: Everolimus-eluting stent
Device: Sirolimus-eluting stent — Sirolimus-eluting stent
  Arms: Sirolimus-eluting stent

SUMMARY:
The purpose of this study is to evaluate whether the newly-approved everolimus-eluting stent is not inferior to the sirolimus-eluting stent in terms of the rate of target-lesion revascularization at 1-year and death or myocardial infarction at 3-year after stent implantation in the real world clinical practice.

DETAILED DESCRIPTION:
Sirolimus-eluting stent is the most widely used coronary drug-eluting stent in Japan. Everolimus-eluting stent is a new coronary drug-eluting stent, which is going to be approved in the first quarter of 2010 by the Japanese Ministry of Health, Labor and Welfare. It has recently been reported that everolimus-eluting stent had lower rate of target-lesion revascularization and stent thrombosis at 1 year as compared with paclitaxel-eluting stent. However, trial results comparing everolimus-eluting stent with sirolimus-eluting stent are largely unknown. The purpose of this study is to evaluate whether the newly-approved everolimus-eluting stent is not inferior to the sirolimus-eluting stent in terms of the rate of target-lesion revascularization at 1-year and death or myocardial infarction at 3-year after stent implantation in the real world clinical practice. The design of this study is all-comer design enrolling patients scheduled for percutaneous coronary intervention using drug-eluting stents without any exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for percutaneous coronary intervention using drug-eluting stents

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3206 (Actual)
Dates: Start 2010-02; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
target-lesion revascularization | 1-year
all-cause death or myocardial infarction | 3-year

SECONDARY OUTCOMES:
all-cause death | 3-year
cardiac death | 3-year
myocardial infarction | 3-year
stent thrombosis (Academic Research Consortium definition) | 3-year
ischemic and hemorrhagic strokes excluding transient ischemic attacks and secondary causes | 3-year
bleeding complications (GUSTO and TIMI definition) | 3-year
stent deployment success | at implantation
procedure time | at implantation
clinically-driven target-lesion revascularization | 3-year
non-target-lesion revascularization | 3-year
coronary artery bypass grafting | 3-year
target-vessel revascularization | 3-year
any repeat coronary revascularization | 3-year
composite of cardiac death, myocardial infarction in the territory of the target vessel or target-lesion revascularization | 3-year
composite of all-cause death, any myocardial infarction or any repeat coronary revascularization | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Shiomi H, Kozuma K, Morimoto T, Kadota K, Tanabe K, Morino Y, Akasaka T, Abe M, Takeji Y, Suwa S, Ito Y, Kobayashi M, Dai K, Nakao K, Tarutani Y, Taniguchi R, Nishikawa H, Yamamoto Y, Nakagawa Y, Ando K, Kobayashi K, Kawai K, Hibi K, Kimura T; RESET Investigators. 7-Year Outcomes of a Randomized Trial Comparing the First-Generation Sirolimus-Eluting Stent Versus the New-Generation Everolimus-Eluting Stent: The RESET Trial. JACC Cardiovasc Interv. 2019 Apr 8;12(7):637-647. doi: 10.1016/j.jcin.2019.01.234. PMID 30947938
- [Derived] Ito S, Watanabe H, Morimoto T, Yoshikawa Y, Shiomi H, Shizuta S, Ono K, Yamaji K, Soga Y, Hyodo M, Shirai S, Ando K, Horiuchi H, Kimura T. Impact of Baseline Thrombocytopenia on Bleeding and Mortality After Percutaneous Coronary Intervention. Am J Cardiol. 2018 Jun 1;121(11):1304-1314. doi: 10.1016/j.amjcard.2018.02.010. Epub 2018 Mar 1. PMID 29628128
- [Derived] Watanabe H, Morimoto T, Shiomi H, Yoshikawa Y, Kato T, Saito N, Shizuta S, Ono K, Yamaji K, Ando K, Kaji S, Furukawa Y, Akao M, Ishikawa T, Tamura T, Yamamoto Y, Muramatsu T, Suwa S, Nakagawa Y, Kadota K, Takatsu Y, Nishikawa H, Hiasa Y, Hayashi Y, Miyazaki S, Kimura T. Mortality impact of post-discharge myocardial infarction size after percutaneous coronary intervention: a patient-level pooled analysis from the 4 large-scale Japanese studies. Cardiovasc Interv Ther. 2019 Jan;34(1):47-58. doi: 10.1007/s12928-018-0517-x. Epub 2018 Mar 5. PMID 29508236
- [Derived] Shiomi H, Kozuma K, Morimoto T, Igarashi K, Kadota K, Tanabe K, Morino Y, Akasaka T, Abe M, Suwa S, Muramatsu T, Kobayashi M, Dai K, Nakao K, Uematsu M, Tarutani Y, Fujii K, Simonton CA, Kimura T; RESET Investigators. Long-term clinical outcomes after everolimus- and sirolimus-eluting coronary stent implantation: final 3-year follow-up of the Randomized Evaluation of Sirolimus-Eluting Versus Everolimus-Eluting Stent Trial. Circ Cardiovasc Interv. 2014 Jun;7(3):343-54. doi: 10.1161/CIRCINTERVENTIONS.113.001322. Epub 2014 May 6. PMID 24803436
- [Derived] Kozuma K, Kimura T, Kadota K, Suwa S, Kimura K, Iwabuchi M, Kawai K, Miyazawa A, Kawamura M, Nakao K, Asano R, Yamamoto T, Suzuki N, Aoki J, Kyono H, Nakazawa G, Tanabe K, Morino Y, Igarashi K. Angiographic findings of everolimus-eluting as compared to sirolimus-eluting stents: angiographic sub-study from the Randomized Evaluation of Sirolimus-eluting versus Everolimus-eluting stent Trial (RESET). Cardiovasc Interv Ther. 2013 Oct;28(4):344-51. doi: 10.1007/s12928-013-0179-7. Epub 2013 Apr 23. PMID 23608784
- [Derived] Kimura T, Morimoto T, Natsuaki M, Shiomi H, Igarashi K, Kadota K, Tanabe K, Morino Y, Akasaka T, Takatsu Y, Nishikawa H, Yamamoto Y, Nakagawa Y, Hayashi Y, Iwabuchi M, Umeda H, Kawai K, Okada H, Kimura K, Simonton CA, Kozuma K; RESET Investigators. Comparison of everolimus-eluting and sirolimus-eluting coronary stents: 1-year outcomes from the Randomized Evaluation of Sirolimus-eluting Versus Everolimus-eluting stent Trial (RESET). Circulation. 2012 Sep 4;126(10):1225-36. doi: 10.1161/CIRCULATIONAHA.112.104059. Epub 2012 Jul 23. PMID 22824435